CLINICAL TRIAL: NCT02713451
Title: Liberal Oxygenation Versus Conservative Oxygenation in Patients With Acute Respiratory Distress Syndrome : Impact on Mortality (LOCO2 Study)
Brief Title: Liberal Oxygenation Versus Conservative Oxygenation in ARDS
Acronym: LOCO2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R/2015/52
Record Dates: First submitted 2016-02-25; First posted 2016-03-18 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2018-11

CONDITIONS: Acute Respiratory Distress Syndrome; Intensive Care
Keywords: Oxygen
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Oxygenation (LO) group (Active Comparator): A modulation of inspired fraction of oxygen will be performed with an objective of PaO2 between 90 to 105 mmHg that will be checked on arterial blood gases (ABG). Between these measurements, SpO2 will be kept more or equal to 96 percent. Alarms will be set at 95 percent for SpO2.
  Interventions: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)
- Conservative Oxygenation (CO) group (Experimental): A modulation of inspired fraction of oxygen will be performed with an objective of PaO2 between 55 to 70 mmHg that will be checked on arterial blood gases. Between these measurements, SpO2 will be kept between 88 and 92 percent. Alarms will be set between 87 and 93 percent for SpO2.
  Interventions: Drug: Modulation of Inspired Fraction of Oxygen (FiO2)

INTERVENTIONS:
Drug: Modulation of Inspired Fraction of Oxygen (FiO2) — In the two groups, if patient is not in the range of arterial oxygen pressure (PaO2), Inspired Fraction of Oxygen (FiO2) will be modified from 5 percent if difference between target is less than 5 mmHg and from 10 percent if difference from target is higher. A new arterial blood gases (ABG) will be performed 30 minutes later to check for the oxygen target range. When ABG are performed, pulsed oxymetry is compared with arterial saturation (SaO2) to adapt survey. Between each ABG, FiO2 is modified from 5 percent to 5 percent each five minutes until reaching good pulsed oxygen saturation (SpO2) target (that can be modified in function of the comparison of arterial oxygen saturation (SaO2 and SpO2 with ABG).
  This management of FiO2 will be done until extubation of the patient.

SUMMARY:
No clear recommendation exists for the level of oxygenation of intensive care patients. In Acute Respiratory Distress Syndrome (ARDS), pulsed oxymetry (SpO2) have to be kept between 88 and 95 percent and oxygen alveolar pressure between 55 and 80 mmHg (PaO2). These recommendations are common but do not lie on high scientific knowledge and level of proof. In the major studies of these fifteen last years that changed ARDS management, PaO2 was kept around 85 and 90 mmHg despite current recommendations of 55 to 80 mmHg of PaO2.

Many recent review and cohort studies pointed the risk of excessive oxygenation especially following cardiac arrest, stroke or traumatic brain injury. However, these data come in majority from cohort or database study without strong definition of hyperoxia. Data coming from prospective studies are scarce and tend to show better outcome of patients with lower objectives of oxygenation in ICU.

High oxygen (O2) level may be deleterious especially on inflammatory lungs. It could enhance injuries due to mechanical ventilation. O2 could be responsable of " hyperoxia induced lung injury ".

The investigators showed in a precedent study that comparing a restrictive oxygenation versus a liberal oxygenation was feasable and do not expose patients to major adverse events. More, mortality at 60 days has tendency to be lower. The investigators therefore ask if a lower objectives of PaO2 in comparison with the level usually seen in last studies on ARDS could improve ARDS patients outcome.

The aim of this study is to show that a restrictive oxygenation in comparison with a liberal oxygenation strategy in patients with ARDS would lower mortality at 28 days.

DETAILED DESCRIPTION:
It is a prospective, comparative, randomized, multicentric, french, open study. Patients with ARDS will be enrolled and will be allocated to Liberal Oxygenation arm (LO) or to Conservative Oxygenation arm (CO) during the invasive mechanical ventilation procedure in ICU.

In LO arm, objective of PaO2 is 90 to 105 mmHg. In CO arm, objective of PaO2 is 55 to 70 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with mechanical ventilation
* ARDS according to Berlin definition:Hypoxemia defined with PaO2 FiO2 ratio less or equal to 300 mmHg with Positive End Expiratory Pressure higher or equal to 5 cmH20, Less than seven days between a known clinical insult or new or worsening of respiratory symptoms, Bilateral opacities on chest Imaging not fully explained by effusions, lobar or lung collapse, or nodules, Respiratory failure not fully explained by cardiac failure or fluid overload
* Less than twelve hours following initiation of mechanical ventilation.

Exclusion Criteria:

* Pregnancy
* Patient less than 18 years old
* Sickle cell disease
* Patient deprived of freedom, Under a legal protective measure
* Cardiac arrest as the reason for ICU hospitalisation
* Traumatic brain injury as the reason for ICU hospitalisation
* Hemoptysis with embolization or surgery
* Extracorporeal life support or Extracorporeal Membrane Oxygenation before randomization
* Chronic Obstructive Pulmonary Disease with oxygen or non invasive ventilation at home (obstructive sleep apnoea syndrome is not an exclusion criteria)
* Patient with very high risk of death with IGS II (Simplified Severity Index II) than 90
* Indication of hyperbaric oxygenation : carbon monoxide intoxication, gas embolism, necrotizing fasciitis
* Cyanide intoxication, methemoglobinemia
* Untreated pneumothorax
* Lymphangitis carcinomatosa
* Eosinophilic pneumonia
* Intensive care management for organ donation
* Participation in another interventional study with mortality as a major outcome to avoid confounding factor
* Patient not affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-28 (Estimated)

PRIMARY OUTCOMES:
Death | Day 28

SECONDARY OUTCOMES:
Death | Day 90
Days free of mechanical ventilation in ICU | Day 28
Sequential Organ Failure Assessment (SOFA) Score | Day 0, 3 and 7
  Sepsis-related Organ Failure Score
Score of morbidity | Day 28
  This score is based on three points: need for mechanical ventilation, need for Morbidity are renal replacement therapy, need of catecholamine or need for ventilation
Ventilator associated pneumonia | Day 28
Septicemia | Day 28
Antibiotic consumption | Day 28
  Number of days exposed to antibiotics divided by the number of days spent in ICU
Cardiovascular complications | Day 28 and day 90
  New onset of rhythm disorders, cardiac ischemia and dose of catecholamin at 28 and 90 days
Neurological evolution | Day 28
  Neurological evolution measured with daily Richmond Agitation Sedation Scale score, seizures, new stroke, daily sedation doses, neuroleptic administration
Respiratory autonomy | Day 28 and 90
  Need for oxygen or mechanical ventilation support

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Barrot, MD, Principal Investigator — BESANCON
Locations (1):
- BARROT Loïc, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Panwar R, Hardie M, Bellomo R, Barrot L, Eastwood GM, Young PJ, Capellier G, Harrigan PW, Bailey M; CLOSE Study Investigators; ANZICS Clinical Trials Group. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Jan 1;193(1):43-51. doi: 10.1164/rccm.201505-1019OC. PMID 26334785
- [Derived] Barrot L, Asfar P, Mauny F, Winiszewski H, Montini F, Badie J, Quenot JP, Pili-Floury S, Bouhemad B, Louis G, Souweine B, Collange O, Pottecher J, Levy B, Puyraveau M, Vettoretti L, Constantin JM, Capellier G; LOCO2 Investigators and REVA Research Network. Liberal or Conservative Oxygen Therapy for Acute Respiratory Distress Syndrome. N Engl J Med. 2020 Mar 12;382(11):999-1008. doi: 10.1056/NEJMoa1916431. PMID 32160661